CLINICAL TRIAL: NCT04865497
Title: A Randomized, Blinded, Single-center, Parallel Controlled , Phase Ⅱ Clinical Trial to Evaluate Immunogenicity and Safety of S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine in Healthy Volunteers Aged From 3 Months to 5 Years Old
Brief Title: Immunogenicity and Safety of S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine in Volunteers Aged From 3 Months to 5 Years Old
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201820301
Record Dates: First submitted 2018-10-15; First posted 2021-04-29 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Dysentery; Dysentery, Bacillary
MeSH Terms: conditions — Dysentery; Dysentery, Bacillary | interventions — HibTITER protein, Haemophilus influenzae

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High dose Group (Experimental): S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine,10μg/dose
  Interventions: Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine; Biological: Haemophilus b Conjugate Vaccine
- Low dose Group (Experimental): S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine,5μg/dose
  Interventions: Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine; Biological: Haemophilus b Conjugate Vaccine
- Adjuvant-free Group (Other): Adjuvant-free S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine,10μg/dose
  Interventions: Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine; Biological: Haemophilus b Conjugate Vaccine
- Control Group (Other): Haemophilus b Conjugate Vaccine,10μg/dose
  Interventions: Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine

INTERVENTIONS:
Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine — Group 1:3/2/1 dose(s) according to age of subjects. Single intramuscular dose contains 10 µg S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine.
  Arms: Adjuvant-free Group; Control Group; Low dose Group
Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine — Group 2:3/2/1 dose(s) according to age of subjects. Single intramuscular dose contains 5 µg S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine.
  Arms: Adjuvant-free Group; Control Group; High dose Group
Biological: S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine — Group 1:3/2/1 dose(s) according to age of subjects. Single intramuscular dose contains 10 µg adjuvant-free S.Flexneriza-S.Sonnei Bivalent Conjugate Vaccine.
  Arms: Control Group; High dose Group; Low dose Group
Biological: Haemophilus b Conjugate Vaccine — Group 1:3/2/1 dose(s) according to age of subjects. Single intramuscular dose contains 10 µg Haemophilus b Conjugate Vaccine.
  Arms: Adjuvant-free Group; High dose Group; Low dose Group

SUMMARY:
The purpose of this study is to evaluate immunogenicity and safety of S.flexneriza-S.sonnei Bivalent Conjugate Vaccine in healthy volunteers aged from 3 months to 5 years old.

ELIGIBILITY:
Inclusion Criteria:

* Health infants and children aged from 3 months to 5 years old.
* Subject or legal representative who consent and has signed written informed consent.
* Subject and parent/guardian who is able to comply with all study procedures.
* Subject who did't receive blood products within 30 days ,immune with any live vaccine within 14 days and inactivated vaccine within 7 days before vaccination.
* Subject who haven't immuned with diarrhea vaccination,3-11 months health infants who haven't immuned with Haemophilus b Conjugate vaccination,or had a history of Hib vaccination before the age of 1 but no history of vaccination after 1 year of age,and the interval between the day of the enrollment and the previous dose is more than one month.
* Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* Febrile illness (temperature ≥ 38°C) in the 3 days or in the acute phase of the disease / active period.
* Subject who have symptoms such as diarrhea, abdominal pain, and pus and bloody stools in the past 3 days.
* Subject who are allergic to tetanus toxoid.
* Allergic history after vaccination.
* Immunodeficiency diseases patients (such as perianal abscess suggests that there may be immunodeficiency in infants and young children) who administered with immunosuppressive agents (≥14 days).
* Subject who are suffering from serious chronic diseases, cardiovascular disease,liver or kidney disease.
* Subject with congenital malformations, drug allergies, convulsions, epilepsy, history of craniocerebral trauma, encephalopathy and psychosis, or family history.
* Subject who diagnosis of thrombocytopenia or other history of coagulopathy may cause intramuscular contraindication.
* Children with abnormal labor（pregnancy week<37w,>42w）,birth weight (<2500g,>4000g), asphyxia rescue history(Only applicable to 3-5 months old group).
* Subject who plan to participate in or is in any other drug clinical trial.
* Any condition that, in the judgment of investigator, may affect trial assessment.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1050 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of adverse events during 30 days | 30 day after each vaccination
  Occurrence of adverse events during a 30 day follow-up period after each vaccination
Antibody positive rate | 30 day after each vaccination
  Percentage of participants with seroresponse to each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Du lin, Master, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Quanzhou Center for Disease Control and Prevention, Quanzhou, Guangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mo Y, Fang W, Li H, Chen J, Hu X, Wang B, Feng Z, Shi H, He Y, Huang D, Mo Z, Ye Q, Du L. Safety and Immunogenicity of a Shigella Bivalent Conjugate Vaccine (ZF0901) in 3-Month- to 5-Year-Old Children in China. Vaccines (Basel). 2021 Dec 28;10(1):33. doi: 10.3390/vaccines10010033. PMID 35062694